CLINICAL TRIAL: NCT06768307
Title: Exploratory Clinical Study of Adebrelimab Combined with Chemotherapy and Concurrent Radiotherapy Versus Sequential Radiotherapy As First-Line Treatment for Extensive-Stage Small Cell Lung Cancer（ES-SCLC）.
Brief Title: Assessment of Adebelizumab Combined with Chemotherapy in Concurrent Radiotherapy Versus Sequential Radiotherapy As First-Line Treatment for Extensive-Stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Rong Yu, MD, Investigator Official Title, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024YJZ108
Record Dates: First submitted 2024-12-23; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: SCLC, Extensive Stage; Immunotherapy; Chemotherapy; Radiotherapy
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: Treatment Protocols for the Two Cohorts drug: Adebrelimab, Carboplatin/Cisplatin, Etoposide
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental): After three cycles of induction therapy with atezolizumab combined with carboplatin/cisplatin plus etoposide, patients who do not show progression will undergo immune-concurrent chemoradiotherapy and immune-sequential chemoradiotherapy, followed by maintenance therapy with atezolizumab until disease progression.
  Interventions: Drug: First-line Immunotherapy Combined with Chemoradiotherapy for ES-SCLC

INTERVENTIONS:
Drug: First-line Immunotherapy Combined with Chemoradiotherapy for ES-SCLC — Cohort 1:
  Induction Phase: Patients will receive three cycles of atezolizumab in combination with carboplatin/cisplatin plus etoposide.
  Concurrent Radiotherapy Phase: the fourth cycle will incorporate concurrent radiotherapy along with atezolizumab and chemotherapy.
  Maintenance Phase: Atezolizumab monotherapy will be administered until disease progression or intolerance by the patient, with atezolizumab being administered for a maximum duration of 2 years.
  Cohort 2:
  Induction Phase: Patients will receive three cycles of atezolizumab in combination with carboplatin/cisplatin plus etoposide.
  Sequential Radiotherapy Phase: the fourth cycle will receive sequential radiotherapy in combination with atezolizumab.Final，Atezolizumab monotherapy will be continued until disease progression.
  Other Names: Adebrelimab

SUMMARY:
Immunotherapy combined with chemotherapy has emerged as the standard of care for patients with extensive-stage small cell lung cancer (ES-SCLC). The incorporation of thoracic radiotherapy can enhance treatment efficacy. Currently, the main types of research investigating immunotherapy combined with thoracic radiotherapy for untreated ES-SCLC are concurrent radiotherapy and sequential radiotherapy. The aim of this study is to evaluate the efficacy of adebelizumab in combination with chemotherapy, when administered concurrently with radiotherapy versus sequentially with radiotherapy, as a first-line treatment for ES-SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, no gender restrictions;
* Confirmed pathological diagnosis of extensive-stage small cell lung cancer (ES-SCLC), defined as disease extending beyond one hemithorax, including malignant pleural and pericardial effusions or hematogenous metastases (according to the Veterans Administration Lung Cancer Study Group, VALG staging); stage IV (any T, any N, M1a/b/c) according to the AJCC (8th edition), or T3-4 due to multiple pulmonary nodules or tumor/nodule size too large to be included in a tolerable radiation therapy plan;
* Participants have not received systemic treatment for extensive-stage SCLC;
* No more than 5 lesions (including metastatic foci), with at least one measurable lesion (according to RECIST v1.1);
* ECOG performance status score of 0-2;
* Life expectancy ≥3 months;
* Consented and signed the informed consent form, willing and able to comply with planned visits, study treatments, laboratory tests, and other trial procedures;
* Normal major organ function, meeting the following criteria (without symptomatic treatment within 14 days): a) Hematology:

Hemoglobin (Hb) ≥90g/L; Platelet (PLT) ≥100×10^9/L; Neutrophil count (ANC) ≥1.5×10^9/L; White blood cell count (WBC) ≥3.0×10^9/L;

Lymphocyte ≥0.5×10^9/L; b) Biochemistry:

Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) ≤ 2.5×ULN; For those with liver metastasis, ALT, AST≤5 ULN; For those with liver or bone metastasis: ALP ≤5 ULN; Total serum bilirubin (TBIL) ≤1.5×ULN (for Gilbert's syndrome participants ≤3×ULN); Albumin (ALB) ≥3 g/dL;

Renal function: Serum creatinine ≤1.5 x ULN or creatinine clearance rate (CrCl) ≥50mL/minute (using Cockcroft/Gault formula); c) Coagulation:

Activated partial thromboplastin time (APTT), International Normalized Ratio (INR), Prothrombin Time (PT) ≤1.5×ULN; d) Others: Lipase ≤1.5 x ULN. Participants with lipase >1.5 x ULN without clinical or radiological evidence of pancreatitis can be included; e) Doppler echocardiography: Left ventricular ejection fraction (LVEF) ≥50%;

* Female participants of childbearing potential must have a negative serum HCG test within 72 hours before the first dose, not breastfeeding, and must use a medically recognized contraceptive method (such as intrauterine devices, birth control pills, or condoms) during the study treatment and for 2 months after the last dose of Adebrelimab or 6 months after the last dose of Carboplatin/Etoposide (whichever is longer); male participants with partners of childbearing potential must be surgically sterilized or agree to use highly effective contraception during the trial and for 2 months after the last dose of Adebrelimab or 3 months after the last dose of Carboplatin/Etoposide (whichever is longer), and no sperm donation during the study.

Exclusion Criteria:

* Participants who have previously received any T-cell co-stimulation or immune checkpoint therapy, including but not limited to cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors, CD137 agonists, or other T-cell targeted drugs.
* Participants who have previously received chemoradiotherapy for limited-stage SCLC;
* Participants with clinically symptomatic central nervous system metastases (such as brain, spinal cord), or leptomeningeal metastases; participants with active or new CNS metastases found on imaging during the screening period are not included. (Asymptomatic untreated CNS metastases with a lesion size <1cm are allowed to be included);
* Participants with multiple liver metastases (isolated liver metastasis participants with metastasis <2cm can be included)
* Participants with spinal cord compression;
* Participants with active autoimmune diseases requiring systemic treatment (such as disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years before the first dose, or with a history of autoimmune diseases and expected recurrence. Replacement therapies (such as thyroid hormone, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic treatment;
* Diagnosed with immune deficiency or receiving systemic glucocorticoid treatment or any other form of immunosuppressive therapy within 14 days before the first dose; the use of physiological doses of glucocorticoids (≤10 mg/day of prednisone or equivalent) is allowed;
* Participants who have had arterial/venous thrombotic events within 6 months before the first dose, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral embolism, etc.), deep vein thrombosis, and pulmonary embolism;
* Participants with a history of idiopathic pulmonary fibrosis, organizing pneumonia (such as cryptogenic organizing pneumonia), drug-induced pneumonia, or idiopathic pneumonia, or evidence of active pneumonia on chest computed tomography (CT) at screening (participants with active tuberculosis are not included);
* Participants who have undergone major surgical treatment or significant traumatic injury within 28 days before the first dose;
* Participants who have received or plan to receive preventive vaccines or live-attenuated vaccines within 4 weeks before the first dose;
* Participants who have received other trial medications or participated in another interventional clinical study within 4 weeks before signing the ICF;
* Participants with other malignancies that require active treatment within 5 years (except for those with a >90% 5-year survival rate such as fully treated basal cell or squamous cell skin cancer, cervical carcinoma in situ, localized prostate cancer after radical surgery, localized bladder cancer, ductal carcinoma in situ after radical surgery, or in situ breast cancer);
* Participants with any severe and/or uncontrolled diseases, including: a) Uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90mmHg) participants; history of hypertensive crisis or hypertensive encephalopathy; b) Uncontrolled cardiac clinical symptoms or diseases such as ≥grade 2 myocardial ischemia or myocardial infarction, uncontrollable arrhythmias (including men QTc ≥450ms, women QTc ≥470ms), and ≥grade 2 congestive heart failure (New York Heart Association, NYHA classification), unstable angina, myocardial infarction within 24 weeks, clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; c) Active or uncontrolled severe infections (≥CTC AE grade 2 infections), including but not limited to hospitalization due to infectious complications, bacteremia, or severe pneumonia, unexplained fever >38.5℃ before the first dose. d) Liver cirrhosis, active hepatitis*; *Active hepatitis - Hepatitis B reference: HBsAg positive, exceeding the upper limit of normal (1000 copies/ml or 500 IU/ml); participants with past Hepatitis B virus (HBV) infection or cured HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HbsAg, and normal HBV DNA values detected during the screening period can be included; *Hepatitis C reference: HCV antibody positive, and HCV viral load exceeds the upper limit of normal/HCV RNA or HCV Ab indicates acute or chronic infection; e) HIV positive or known Acquired Immune Deficiency Syndrome (AIDS); f) Urine routine suggests urinary protein ≥++, and confirmed 24-hour urinary protein quantification >1.0 g;
* Participants with clinically symptomatic third-space fluid accumulation, such as pericardial effusion, pleural effusion, and abdominal effusion requiring repeated drainage (such as once a month or more frequently) that cannot be controlled by tapping or other treatments;
* Participants whose adverse events (except for alopecia) caused by previous treatments have not recovered to ≤CTCAE grade 1; other toxicities caused by previous antitumor treatments that are expected to be unresolved and have long-term persistent sequelae, such as neurotoxicity caused by platinum-based treatments, are allowed to be included;
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* Known history of drug abuse that cannot be quit, mental disorders, alcoholism, drug abuse, or substance abuse;
* Known allergy to study drugs or excipients, known severe allergic reactions to any monoclonal antibody;
* As judged by the investigator, there are factors that seriously endanger the safety of the participants or other factors that may lead to the forced termination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From enrollment to the end of treatment at 1 year
  From the date of enrollment to the date of disease progression

SECONDARY OUTCOMES:
OS | From date of enrollment to maximum of 2 years or death
  from the date of enrollment until death by any cause or last follow-up
Treatment-related adverse events | Duration of treatment and follow up until death or 90 days after enrollment
  Treatment-related adverse events according to CTCAE 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes